CLINICAL TRIAL: NCT01512810
Title: Treatment of Endometrial Cancer Utilizing Pathology Intraoperative Consultation to Determine Extent of Surgical Staging
Brief Title: Intraoperative Pathological Evaluation for Surgical Treatment & Staging for Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Frederick R. Ueland, M.D. (Other)
Responsible Party: Sponsor-Investigator, Frederick R. Ueland, M.D., Professor, Obstetrics and Gynecology, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-GYN-130
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Endometrial Cancer
Keywords: Endometrial; Cancer; Intraoperative Consultation
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms | interventions — Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-risk for nodal involvement (No Intervention): No lymphadenectomy recommended
- High-risk for nodal involvement (Experimental): Lymphadenectomy recommended, including: obturator, iliac (internal, external, common) and aortic lymph nodes
  Interventions: Procedure: Lymphadenectomy

INTERVENTIONS:
Procedure: Lymphadenectomy — Lymphadenectomy recommended, including: obturator, iliac (internal, external, common) and aortic lymph nodes
  Arms: High-risk for nodal involvement

SUMMARY:
Complete pelvic and para-aortic lymphadenectomy performed at the time of primary surgical staging for endometrial cancer increases operative time and surgical morbidity, but appears to be necessary in most high grade and deeply invasive cancers. To date, the Mayo Clinic approach has not been reproduced, and the investigators propose to validate their algorithm at the University of Kentucky utilizing intra-operative consultation (IOC). The preliminary data at the University of Kentucky for IOC and endometrial cancer outcomes suggest that the investigators are well-suited to perform this investigation. A surgical approach that is tailored to the patient's cancer biology is rational, supported by the recent literature, and medically compelling since the co-morbidities of many obese, low-risk EC patients put them at significantly increased perioperative risk for complete lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be surgical candidates for complete hysterectomy and bilateral salpingo-oophorectomy and pelvic and aortic lymphadenectomy.
* Patients must have a histologically confirmed diagnosis of endometrial cancer and no clinical evidence of extra-uterine disease on preoperative evaluation.
* Preoperative evaluation to rule-out extra-uterine disease may include CT scan, MRI, or ultrasound. Preoperative imaging is not mandatory for study enrollment.
* Patients may have received prior systemic chemotherapy. Such therapy must have been completed at least 5 years prior to study entry and the patient has no evidence of disease subsequent to such therapy. Patients must not have received neoadjuvant chemotherapy for the present disease.
* Patients must have GOG performance status 0, 1, or 2.
* Patients must have an estimated survival greater than or equal to 3 months
* Patients who have met the pre-entry requirements specified in Section 7.0.
* Patients must have signed an approved informed consent and HIPAA authorization.

Exclusion Criteria:

* Patients with clinical evidence of disease beyond the uterus, including presence of suspicious aortic or inguinal nodes on imaging or clinical exam.
* Patients who have received previous vaginal, pelvic, or abdominal irradiation.
* Patients who received chemotherapy directed at the present disease.
* Patients who have circumstances that will not permit completion of this study or the required follow-up.
* Patients with renal abnormalities, such as pelvic kidney, horseshoe kidney, or renal transplantation, that would require modification of surgical lymph node assessments.
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer within the last five years.
* Patients with GOG Performance Grade of 3 or 4.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival | 24 months
  Recurrence-free survival rates in low-risk and high-risk subgroups of patients with endometrial cancer as classified by the use of pathology intraoperative consultation (IOC).

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Ueland, M.D., Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No